CLINICAL TRIAL: NCT01220310
Title: Doctors and Web-based Self-management Support Pilot Study.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other); Alameda County Medical Center (Other)
Responsible Party: Principal Investigator, Kate Lorig, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SU-09242008-1309; IRB Protocol ID: 15108
Record Dates: First submitted 2010-08-12; First posted 2010-10-13 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Online diabetes workshop observation and learning sessions
  Interventions: Behavioral: Online diabetes workshop observation and learning sessions

INTERVENTIONS:
Behavioral: Online diabetes workshop observation and learning sessions — We will, by self-administered pre- and post-intervention surveys, evaluate the effectiveness of the online diabetes workshop observations and learning sessions.

SUMMARY:
Doctors and web-based self-management support pilot study will test whether health professionals' observation of an online patient workshop on self-management of diabetes and participation in structured learning sessions on self-management strategies will change the attitudes and confidence of physicians and other health professionals regarding their willingness and ability to perform self-management interventions with patients. If this pilot suggests that attitudes and confidence levels can change, we hope to launch a larger study to examine this method of learning and its effectiveness in more detail.

DETAILED DESCRIPTION:
The standard of care is that health professionals receive their usual education on self-management, which ranges from minimal to modest, depending on the training site. They will be identified and invited to attend by the program director and/or clinic managers.

Health professional participants will attend 60-90 minutes teaching sessions with other health professionals, either in person or via Web-Ex, once per week for a total of 4 weeks. The program director and/or clinic managers overseeing these health professionals will make room for these sessions in their clinic schedule, so that you have no clinical or other responsibilities during those times.

During the first session, the Principal Investigator will first read the informed consent/fact sheet to the health professionals and ask for any questions. A copy of the informed consent/fact sheet will be given to each health professional participant, and they will be asked to provide their contact information on a sign up sheet. At that point, they will complete their first survey questionnaire.

Between these group sessions, at the convenience of the participant, the health professional will log-on to the online workshop to observe the patients' progress in the online course. The health professional will be expected to log on 3 times per week for approximately 10 minutes at a time. The health professional will have 2 'homework' assignments during the entire 4 weeks of learning sessions. These consist of thinking critically about how the self-management techniques they observe patients using online might apply to other patients the health professionals observe, whether online or in their clinics.

The health professionals will also be asked to complete voluntary pre- and post-course surveys. There will be time set aside during the first and last learning sessions for them to complete the surveys.

The final learning session will primarily be devoted to a focus group discussion of the learning sessions. The total time commitment to the observational learning sessions is to attend the 4 learning sessions (60-90 minutes apiece once per week), visit the patient online workshop site 3 times per week (for at least 10 minutes a time), and do the 'homework' assignments (which are expected to take 10-20 minutes apiece to complete).

The health professionals will not actually participate in the online workshop for patients. In fact, if they decide to participate in this project, they are instructed not interact in any way with the patients in the online workshop. The health professionals must agree to observe only, not to post on the discussion boards, and not to answer any messages that they may receive via the online messaging system. The workshops are monitored by Stanford staff, and they will take any action necessary if the health professionals alert them to the need to respond to a patient.

ELIGIBILITY:
Inclusion Criteria:Health professional at primary care clinic of participating site identified by their residency director and/or clinic manager as having the schedule flexibility to attend (convenience sample). Can include physicians (residents and attendings), registered nurses, medical assistants, dieticians, community health workers, and the like. In the case of the residents, they will be on outpatient clinic blocks for the month of the learning sessions, and the program directors have the ability to free up their schedules to allow for participation in the learning sessions. Exclusion Criteria:The health professionals that do not want to participate, or are not working at one of partner sites, or the residency director and/or clinic manager determines that the health professional's schedule does not have the flexibility in it to allow for regular participation in the learning sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Alameda County Medical Center, Oakland, California
  - O'Connor Hospital, San Jose, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California